CLINICAL TRIAL: NCT05575674
Title: Retrospective Study on Myoelectric Elbow-Wrist-Hand Orthosis User Outcomes During Home Use
Brief Title: Retrospective Study on Myoelectric Elbow-Wrist-Hand Orthosis User Outcomes
Status: Completed | Type: Observational
Sponsor: Myomo (Industry)
Collaborators: Orthocare Innovations, LLC (Industry); Geauga Rehabilitation Engineering, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: PRO-002
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Brachial Plexus Injury; Spinal Cord Injuries; Neurological Disease
Keywords: MyoPro
MeSH Terms: conditions — Stroke; Spinal Cord Injuries; Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Myoelectric Elbow-Wrist-Hand Orthosis — An arm orthosis that uses myoelectric signals to control the level of mechanical assistance provided to a user's elbow and hand in order to overcome upper limb weakness or paralysis and achieve functional tasks.
  Other Names: MyoPro®

SUMMARY:
The objective of this study is to retrospectively evaluate the outcomes and clinical benefits provided by this brace to adult patients with upper limb impairment or paralysis due to brachial plexus, stroke (CVA), spinal cord injury, or other neurological disease or injury.

DETAILED DESCRIPTION:
The objective of this study is to retrospectively evaluate the outcomes and clinical benefits provided by this brace to adult patients with upper limb impairment or paralysis due to brachial plexus, stroke (CVA), spinal cord injury, or other neurological disease or injury.

The primary result in this study is a comparison of the Disabilities of the Arm, Shoulder and Hand questionnaire results that were completed before and at least six months after receiving the MyoPro. A retrospective record review will be done to collect data regarding MyoPro user outcomes for individuals that received a MyoPro starting January 2021 and after. Additional data types such as demographics and clinical outcomes will be gathered. Participants may complete at least one follow-up session to record responses to additional inquiries from the research team.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 65 years and older at the time of MyoPro delivery
* Completed the DASH questionnaire at evaluation before receiving the MyoPro
* Completed the DASH questionnaire at least six months after receiving the MyoPro
* Has intact cognition
* Able to clearly and verbally communicate in the English language

Exclusion Criteria:

* Life-changing event(s) or change(s) in medical status that affected ability to use the MyoPro
* Did not complete the DASH after receiving the MyoPro
* Other conditions (e.g., cognitive issues) or circumstances that would preclude safe and/or effective participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adult with upper limb impairment caused by brachial plexus injury, stroke, or spinal cord injury, or other neurological disease or injury who have been fitted with a myoelectric Elbow-Wrist-Hand orthosis.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) | Pre-MyoPro
  Validated outcome measure that asks an individual to self-report about the ability to perform certain upper limb activities. Questions are responded on a 5-point Likert scale.
Disabilities of the Arm, Shoulder and Hand (DASH) | At least six months Post-MyoPro
  Validated outcome measure that asks an individual to self-report about the ability to perform certain upper limb activities. Questions are responded on a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Chang, Principal Investigator — Orthocare Innovations, LLC
Locations (3):
- United States (3):
  - Myomo, Inc., Boston, Massachusetts
  - Geauga Rehabilitation Engineering, Inc., Chardon, Ohio
  - Orthocare Innovations, LLC, Edmonds, Washington

IPD SHARING:
Plan to Share IPD: No